CLINICAL TRIAL: NCT00002262
Title: A Phase I/II Study of Intralesional Recombinant Tumor Necrosis Factor in Patients With AIDS-Related Cutaneous Kaposi's Sarcoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 066A; 86-989
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1988-12

CONDITIONS: Sarcoma, Kaposi; HIV Infections
Keywords: Skin Neoplasms; Tumor Necrosis Factor; Acquired Immunodeficiency Syndrome
MeSH Terms: conditions — Sarcoma, Kaposi; HIV Infections; Skin Neoplasms; Acquired Immunodeficiency Syndrome | interventions — Tumor Necrosis Factor-alpha

INTERVENTIONS:
Drug: Tumor Necrosis Factor

SUMMARY:
To evaluate tolerance, toxicity, and preliminary evidence of antitumor efficacy of intralesionally administered tumor necrosis factor (TNF) and to define a maximum tolerated dose (MTD) for single intralesional injections. In addition, to assess the effects of TNF injections on Kaposi's sarcoma (KS) lesions as measured by P-32 magnetic resonance spectroscopy.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* Biopsy-proven Kaposi's sarcoma (KS) with multiple cutaneous lesions.
* Minimum life expectancy of 3 months.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* Clinically significant cardiac disease.
* Known hemorrhagic diathesis or active bleeding disorder.
* Clinically apparent vascular disease.
* Known lipoprotein disorders.
* History of seizure disorder or central nervous system (CNS) metastasis.
* Additional malignancy.

Concurrent Medication:

Excluded:

* Cardiac agents.
* Anticoagulants.
* Thrombolytic agents.
* Nonsteroidal anti-inflammatory drugs.
* Corticosteroids.
* Aspirin.
* Vasodilators.

Patients with the following are excluded:

* Additional malignancies or other conditions listed in Patient Exclusion Co-Existing Conditions.

Prior Treatment:

Excluded within 4 weeks of study entry:

* Chemotherapy.
* Radiotherapy.
* Immunotherapy.

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- San Francisco AIDS Clinic / San Francisco Gen Hosp, San Francisco, California, United States